CLINICAL TRIAL: NCT04857216
Title: Comparison of the Block Characteristics of Ultrasound Guided Costoclavicular and Infraclavicular Block With the Perfusion Index
Brief Title: Comparison of the Block Characteristics of USG Guided Costoclavicular and Infraclavicular Block With the Perfusion Index
Status: Completed | Type: Observational
Sponsor: Izmir Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Arslan Yurtlu, Associate Professor, Izmir Ataturk Training and Research Hospital
Other Study IDs: IATRH
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Costoclavicular and Infraclavicular Block for Patients Who Have Undergone Hand,Forearm and Arm Surgery
Keywords: infraclavicular, costoclavicular, perfusion index, block
MeSH Terms: conditions — Bites and Stings | interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infraclavicular Group: Block Characteristics of Ultrasound Guided Infraclavicular Block with the Perfusion Index
  Interventions: Device: Perfusion Index
- Costoclavicular Group: Block Characteristics of Ultrasound Guided costoclavicular Block with the Perfusion Index
  Interventions: Device: Perfusion Index

INTERVENTIONS:
Device: Perfusion Index — perfusion index in the prediction of peripheral block success was previously reported for infraclavicular brachial plexus block, axillary brachial plexus block, interscalene brachial plexus block, and supraclavicular brachial plexus in adult patients

SUMMARY:
With this study, it was aimed to compare the block characteristics evaluated with traditional methods in infraclavicular and costoclavicular block applications performed in upper extremity surgery in our clinic with the perfusion index

DETAILED DESCRIPTION:
Peripheral nerve block is to anesthetize the dermatomes belonging to the nerve or nerve group to which the block is applied, by performing sympathetic, sensory and motor blocks. Brachial plexus blockade; It is a peripheral nerve blockage that can be used in surgical operations to be performed on the upper extremity and can be performed at the level of interscalene, supraclavicular, infraclavicular, costoclavicular, axillary and terminal nerves.

The costoclavicular brachial plexus block has been used as an alternative to lateral sagittal infraclavicular block, due to its ease of application, its rapid onset of action and its high success rate. The effectiveness of the block is measured by sensory, motor and sympathetic block effects. The sensory block can be evaluated by cold or pinprick test, and motor block by traditional methods such as the patient's response to verbal commands and can be objective.

Sympathetic block manifests itself with vasodilation and an increase in blood flow rate and can be measured with the more quantitative perfusion index (PI). The perfusion index represents the ratio of pulsatile blood flow to static blood flow in peripheral tissue and can be measured continuously and noninvasively from a pulse oximeter. Successful peripheral nerve blockade; It is seen as local vasodilation, increased local blood flow, some increase in skin temperature and loss of sensation in the extremity due to the blockage of sympathetic fibers. It can be a guide in determining the effectiveness of the block because it is noninvasive and easy, providing rapid evaluation, without requiring patient cooperation to evaluate the success of the block.

ELIGIBILITY:
Inclusion Criteria:

* All costoclavicular and infraclavicular block patients who have undergone hand,forearm and arm surgery
* Patients over the age of 18

Exclusion Criteria:

* Patients who do not want to participate in the study
* Patients whose peripheral block administration is contraindicated

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All costoclavicular and infraclavicular block patients who have undergone hand,forearm and arm surgery over the age of 18
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Correlation of perfusion index with infraclavicular and costoclavicular block success | 3 Months
  Correlation of perfusion index with infraclavicular and costoclavicular block success

SECONDARY OUTCOMES:
Comparison of the Block Characteristics of Ultrasound Guided Costoclavicular and Infraclavicular Block | 3 Months
  Comparison of the Block Characteristics of Ultrasound Guided Costoclavicular and Infraclavicular Block

CONTACTS AND LOCATIONS:
Overall Officials: Busra Serce, MD, Study Director — KCU Izmir Atatürk Training And Research Hospital; Derya Yurtlu, MD, Principal Investigator — KCU Izmir Atatürk Training And Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Katip Celebi University Atatürk Training and Research Hospital, Izmir
  - Katip Çelebi University İzmir Atatürk Training and Reseach Hospital, Izmir